CLINICAL TRIAL: NCT05832957
Title: The Effectiveness of Cognitive-Functional Intervention to Reduce Driving Risk Factors of Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Navah Ratzon, Head of Health Professions, Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anat Keren
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Driving Risk Factors Among Adolescents With ADHD
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drive fun (Experimental): The intervention will include 11 sessions and last 11-13 weeks. Seven intervention meetings will be individual sessions of one hour at the driving lab at Tel Aviv University and four 90-minute meetings will be group sessions (3-6 participants) and will be conducted remotely by Zoom. The parents will be present during the first and last individual sessions
  Interventions: Behavioral: Drive fun
- educational intervention (Experimental): 7 individual sessions of one hour at the driving lab at Tel Aviv university and 4 group sessions- 90 minutes by Zoom of group sessions of an educational intervention of safe driving according to Ministry of Education. The intervention focuses only on the cognitive aspects since it is based on imparting educational knowledge regarding safe driving with opportunities for gamified, non-driving-related activities such as board games (e.g., rush hour) and social games
  Interventions: Behavioral: educational intervention
- No Intervention (Other): one-time short guidance on safe driving at the end of the study.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Drive fun — The "Drive Fun" intervention program aims to promote the development of adaptive self-awareness and facilitate the acquisition of management strategies that foster safe and confident driving among participants. The program utilizes a driving simulator to provide a guided learning experience, which incorporates various sources of information, as well as games and thinking tasks. Additionally, participants will engage in reflective exercises that draw upon their occupational experiences and their driving performance within the simulator. Parental involvement is also incorporated to ensure ongoing support for the continued practice of learned skills.
  Arms: Drive fun
Behavioral: educational intervention — 7 individual sessions of one hour at the driving lab at Tel Aviv university and 4 group sessions- 90 minutes by Zoom of group sessions of an educational intervention of safe driving according to Ministry of Education. The intervention focuses only on the cognitive aspects since it is based on imparting educational knowledge regarding safe driving with opportunities for gamified, non-driving-related activities such as board games (e.g., rush hour) and social games
  Arms: educational intervention
Other: No intervention — one-time short guidance on safe driving at the end of the study.
  Arms: No Intervention

SUMMARY:
Background: Attention deficit hyperactivity disorder (ADHD) is associated with a high risk for driving accidents. Adolescents with ADHD are 1.2 to 4 times more prone to be involved in car accidents. Driving accidents are the leading cause of death among adolescents.

Objective: Examining a multidimensional applied intervention based on serious gaming principles to improve the driving capabilities and skills of adolescents with ADHD Methodology: The study will include 90 adolescents (aged 15-18 years old) with ADHD diagnosis who did not yet start driving lessons. Participants will undergo a stratified randomized clinical trial, single-blinded. The stratified randomization process will include gender, age, and medication status. There exist three different intervention modalities: (1) A personalized cognitive-functional intervention- 'Drive-Fun' (group1) (2) educational intervention (group2); and (3) no intervention (group3). Meetings will entail 11 once-a-week sessions. Participants will be evaluated before intervention (baseline), after the intervention, and at a 6-month follow-up. Evaluations will include simulated driving skills, meta-cognitive abilities, eye tracking, and brain activity (EEG) measures. The evaluation and the intervention will be conducted by two certified occupational therapists. Participants and the therapist performing the evaluations will be blinded to group type and intervention.

The potential scientific contribution of the proposed research: Given the great risks of injury to adolescents with ADHD and other road users, it is important to identify dangerous driving behaviors as well as develop methods that can lead to better driving skills and a safer driving experience. It is anticipated that evidence will be presented by the evaluation battery that the personalized intervention program developed will significantly improve potential driving skills on the simulator and hopefully also actual driving.

DETAILED DESCRIPTION:
Background: Attention deficit hyperactivity disorder (ADHD) is associated with a high risk for driving accidents. Adolescents with ADHD are 1.2 to 4 times more prone to be involved in car accidents. Driving accidents are the leading cause of death among adolescents.

Objective: Examining a multidimensional applied intervention based on serious gaming principles to improve the driving capabilities and skills of adolescents with ADHD Methodology: The study will include 90 adolescents (aged 15-18 years old) with ADHD diagnosis who did not yet start driving lessons. Participants will undergo a stratified randomized clinical trial, single-blinded. The stratified randomization process will include gender, age, and medication status. There exist three different intervention modalities: (1) A personalized cognitive-functional intervention- 'Drive-Fun' (group1) (2) educational intervention (group2); and (3) no intervention (group3). Meetings will entail 11 once-a-week sessions. Participants will be evaluated before intervention (baseline), after the intervention, and at a 6-month follow-up. Evaluations will include simulated driving skills, meta-cognitive abilities, eye tracking, and brain activity (EEG) measures. The evaluation and the intervention will be conducted by two certified occupational therapists. Participants and the therapist performing the evaluations will be blinded to group type and intervention.

The potential scientific contribution of the proposed research: Given the great risks of injury to adolescents with ADHD and other road users, it is important to identify dangerous driving behaviors as well as develop methods that can lead to better driving skills and a safer driving experience. It is anticipated that evidence will be presented by the evaluation battery that the personalized intervention program developed will significantly improve potential driving skills on the simulator and hopefully also actual driving.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD by a psychiatrist according to DSM -V
* Did not begin driving lessons.

Exclusion Criteria:

A chronic primary psychiatric diagnosis A primary developmental disorder that is not ADHD (e.g., Autism Spectrum Disorder).

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-02-10 (Actual); Study Completion 2026-02-10 (Actual)

PRIMARY OUTCOMES:
Reducing errors while driving on a driving simulator | 1 year
  The expectation is that the subjects will drive better and their simulation will have fewer mistakes such as going through a red light or driving at excessive speed

CONTACTS AND LOCATIONS:
Locations (1):
- ; The faculty of medicine & health professions, Tel-Aviv University,, Tel Aviv, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No